CLINICAL TRIAL: NCT03378167
Title: PediCRaFT: Pediatric Crohn's Disease Fecal Microbiota Transplant Pilot Study
Brief Title: PediCRaFT: Pediatric Crohn's Disease Fecal Transplant Trial
Acronym: PediCRaFT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster Children's Hospital (Other)
Collaborators: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Nikhil Pai, Associate Professor, Division of Pediatric Gastroenterology & Nutrition, McMaster Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0000
Record Dates: First submitted 2017-12-12; First posted 2017-12-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Crohn Disease; Pediatric Crohns Disease; Inflammatory Bowel Diseases; Colitis
Keywords: Paediatrics; Pediatrics; Crohn's; Crohn; Microbiome; Microbiota; FMT; Fecal Transplant; Fecal Microbiota Transplant; IBD-U; Inflammatory Bowel Disease Unclassified; Inflammatory Bowel Disease Indeterminate; IBD; Colitis
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Colitis | interventions — Microbiota; Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 2:1 to one of two groups upon consent: intervention or control. 30 patients will be randomized to receive an FMT via colonoscopy + oral microbiota capsular (OMC) therapy (INTERVENTION), and 15 patients will be randomized to receive normal saline (NS) via colonoscopy + dextrose-containing oral capsules (oral placebo capsule, OPC) (CONTROL). Randomization will occur through a computer-generated block-randomization pattern (block size = 6 participants).
  Patients randomized to the control group will be given the option of receiving open-label treatment, with the intervention therapy, either: upon completion of the trial, or if they are removed from the trial due to disease exacerbation or other adverse event, at the discretion of their primary gastroenterologist.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: COLONOSCOPY:
  1. Microbial enemas are drawn up in a 500cc syringe that is concealed with an opaque bag, used to infuse contents through the colonoscope. This will insure contents are blinded to non-study personnel in the room
  2. Patients randomized to the control study arm will have identical concealment of the 500cc syringe used to infuse contents through the colonoscope. For the NS infusion, study personnel will add an additional 0.75 ml of commercially available (Club House® brand), food-grade food coloring (2 drops red, 3 drops green, 7 drops yellow) to confer a brown color to the clear normal saline solution. This step will maintain blinding for the patient and non-study personnel in the room, as the contents of the liquid will be visible endoscopically, but will still retain a similarly-colored brown appearance akin to human stool.
  ORAL CAPSULAR THERAPY:
  a), b) The opaque color of both the OMC and OPC will insure that blinding is preserved to the study patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MICROBIOTA (Experimental): Patients randomized to the INTERVENTION arm will receive a baseline fecal microbiota transplant (FMT) colonoscopic infusion at Week 0, followed by twice-weekly oral microbiota capsule (OMC) therapy for 6 weeks (including Week 0). (n = 30)
  Interventions: Biological: MICROBIOTA
- PLACEBO (Placebo Comparator): Patients randomized to the CONTROL arm will receive a baseline normal saline (NS) colonoscopic infusion at Week 0, followed by twice-weekly dextrose-containing oral placebo capsule (OPC) therapy for 6 weeks (including Week 0). (n = 15)
  Interventions: Biological: PLACEBO

INTERVENTIONS:
Biological: MICROBIOTA — Fecal microbiota enema (RBX2660) infused via colonoscope x 1 + oral microbiota capsules (RBX7455) x 6 weeks. The fecal microbiota enema (RBX2660) prepared by Rebiotix has received Health Canada Clinical Trials Application (CTA), and U.S. Food and Drug Administration Investigational New Drug Application (IND) approval for clinical trials in patients with recurrent Clostridium difficile infection, and pediatric inflammatory bowel disease. The human-derived fecal oral microbiota capsule (RBX7455) has received U.S. Food and Drug Administration Investigational New Drug Application (IND) approval for clinical trials in patients with recurrent Clostridium difficile infection.
  Other Names: RBX2660; RBX7455; Fecal microbiota transplant
  Arms: MICROBIOTA
Biological: PLACEBO — Placebo enema (Normal Saline) infused via colonoscope x 1 + oral placebo capsules (dextrose-containing capsules) x 6 weeks.
  NOTE: Patients randomized to the control group will be given the option of receiving open-label treatment, with the intervention therapy, either: upon completion of the trial, or if they are removed from the trial due to disease exacerbation or other adverse event, at the discretion of their primary gastroenterologist.
  Arms: PLACEBO

SUMMARY:
The objective of this study is to assess the feasibility of a novel colonic and oral fecal microbiota transplantation protocol for the treatment of active pediatric Crohn's disease (CD). Specifically, we will test the hypothesis that a protocol of combination fecal microbiota colonoscopic infusion and oral microbiota capsules (OMC), using live fecal material from anonymous unrelated donors, can improve the disease activity of pediatric CD patients.

DETAILED DESCRIPTION:
Several recent studies have assessed the role of fecal microbiota transplantation (FMT) in the treatment of inflammatory bowel disease (IBD). IBD is a chronic autoimmune gastrointestinal disorder that has been associated with disease-specific microbial signatures in the host. The vast majority of literature on the therapeutic role of FMT has assessed its role in the treatment of acute Clostridium difficile colitis, but its effectiveness at treating this disease condition suggests a central role of the microbiome in host immune tolerance.

A. Alterations in the IBD Microbiome Investigators have characterized specific alterations of the gut microbiota in ulcerative colitis and Crohn's disease, compared to healthy controls. Patients with active IBD may have a relative depletion in anaerobic microbes, such as Bacteroides vulgatus, Lachnospiraceae (p: Firmicutes), and an increase in Proteobacteria and Bacillus (p: Firmicutes). These microbial signatures of IBD have led to several hypotheses about the protective, and pathological roles of different resident intestinal bacterial species. Conte et al have suggested that B. vulgatus may have a protective role against colitis, downregulating inflammation. Other studies have suggested that dysbiosis in IBD leads to decreased production of key short-chain fatty acids, such as butyric acid metabolized by Faecalibacterium prausnitzii. Directly, butyric acid and other short-chain fatty acids are key substrates absorbed by colonocytes, and indirectly, butyrate may inhibit inflammatory processes in the intestinal mucosa by suppressing cytokines, like interleukin-8. These studies have attempted to define canonical "intestinal-microbial-immune axes," supporting the hypothesis that IBD may occur secondary to an altered microbiome in a genetically, immunologically susceptible host. This constant host-microbial cross-talk may thus be altered by the introduction of key bacterial species that are otherwise absent, or decreased as a consequence of active mucosal inflammation, in the IBD gut. While FMT would not provide targeted, species-specific inoculations, whole stool transplant would theoretically introduce a broad range of bacteria, including those that are theoretically "favorable" to the host.

B. The Pediatric Microbiome Pediatric IBD, and the pediatric microbiome, have several unique features that suggest microbial-based therapies could be particularly effective. Crohn's disease and ulcerative colitis typically have a much more aggressive course in the pediatric age group, suggesting that the pediatric IBD phenotype may have a pathophysiology that is distinct from adult-onset IBD. In pediatric IBD, the early age of onset makes the cumulative burden of medications, nutritional impairment, and surgery greater. Several standard IBD medication therapies have unique, age-specific toxicities in children. The overlap of pediatric chronic disease with critical periods of growth, bone accretion, and psychosocial development can make disease exacerbations disproportionately affect a child's long-term outcome. The pediatric microbiome itself has key differences. The shorter latency of disease may offer a unique window to reverse an underlying state of "dysbiosis." The pediatric microbiome may be more malleable than a fully defined adult microbiome, and the relatively immature immune system of children may be more influenced by FMT.

C. FMT for the Treatment of Pediatric IBD Four case series have been published for the treatment of pediatric ulcerative colitis (UC) and CD using FMT. Protocols varied between all studies, and three main routes of administration were used: serial enemas, serial enemas with supplementary colonoscopic administration, and nasogastric tube. The first published study, involved five enemas administered daily to 9 UC patients, ages 7-21. Outcomes included clinical improvement from baseline using Pediatric Ulcerative Colitis Activity Index (PUCAI) scores, at one-week, and one-month post-treatment. 6/9 patients maintained clinical response at their one-month follow-up assessment. In 2015, two case series of FMT for CD and UC patients were published. A single FMT infusion was administered via nasogastric tube (NGT) to 4 UC, and 9 CD patients. No clinical response was seen in UC through NGT administration. In contrast, remission was induced in 7/9 CD patients within 2-weeks post-treatment, with 5/9 maintaining remission at week 6 and week 12. The most recent pediatric case series from 2015 included a cohort of pediatric UC patients treated with oral 5-ASA monotherapy, who received a combination of serial FMT enemas and colonoscopic infusions. 3 patients were included; 100% went into clinical remission at week 2, sustained clinical remission at week 4, and had complete withdrawal of immunotherapy at time of publication. Within the limitations of this small case series, there was a correlation between the number of FMT administrations, and the duration of remission.

Two single-center pediatric case reports have recently been published showing marked clinical improvement in two patients with severe colitis. A 2015 case report describes a 4-month old female presenting with an early-onset colitis with UC-like phenotype. The patient was refractory to treatment with azathioprine and corticosteroids, and did not respond to further treatment with probiotics, a trial of amino-acid based formula, or infliximab. 2 serial FMT infusions with anonymous donor stool were administered via colonoscope, and a subsequent 5 infusions via nasoduodenal tube. These interventions led to clinical improvement, and complete resolution of histopathologic changes 6-months post FMT. A recent, 2016 case report describes an 11-year old female with corticosteroid-dependent UC who was unresponsive to treatment with 5-aminosalicylic acid and tacrolimus14. An initial FMT using her father's donor stool was performed via colonoscopy, and subsequent daily FMTs via fecal retention enema over the next 4 days, followed by 11 additional FMTs via retention enema every 2 to 4 weeks over 10 months. The patient remained in clinical remission at 40 weeks post final FMT, and showed complete endoscopic healing.

D. Clinical Observations from Published Pediatric IBD FMT Studies Despite promising results, major drawbacks to these four pediatric studies include small sample sizes and their open label study design. Studies of clinical response demand a blinded study protocol, particularly given that many patients who enrol in FMT studies are a self-selected group, who already believe in the therapeutic value of "natural" treatments. Further, inflammatory bowel disease has well-described associations between clinical symptoms, mucosal disease activity and underlying stressors; thus, patient bias may have a significant influence on self-reported PUCAI/PCDAI (Pediatric Crohn's Disease Activity Index) scores when measuring clinical response. In addition, it is also important to note that success of FMT for IBD reflected in the aforementioned studies may reflect a propensity for studies with positive results to be published and unreported, unsuccessful studies may exist.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients
* ≥3yo
* Crohn's disease, or IBD-Unclassified favoring Crohn's disease (as deemed by the patient's primary pediatric gastroenterologist)
* Active symptoms

Exclusion Criteria:

* Currently enrolled in another clinical trial
* Unable to give informed consent or assent
* Severe comorbid medical illness (at discretion of patient's primary pediatric gastroenterologist)
* Concomitant Clostridium difficile infection
* Severe Crohn's disease flare requiring hospitalization
* Commenced new, or temporary medical therapies (ie. corticosteroids, antibiotics, prebiotics) within 4 weeks prior to commencing the trial; NB: Weaning doses of corticosteroid will be permitted (≤ 0.25mg/kg/day)

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Monthly Recruitment Rate | 30 weeks
  Assessment of recruitment rate (based on patients meeting all eligibility criteria who were approached for trial entry)
Dropout Rate Post Enrolment | 30 weeks
  Rate of patients leaving the trial (patient, or protocol directed exclusion) after enrolment
Rate of Patient Protocol Adherence | 30 weeks
  Rate of patients providing all required blood, stool and urine samples per protocol
Rate of Adverse Events | 30 weeks
  Rate of patients requiring hospitalization, or experiencing PCDAI increase ≥20 x 2 successive measures

SECONDARY OUTCOMES:
Clinical: Improvement in Disease Symptoms | Baseline, Week 6, Week 30
  PCDAI decrease ≥15 from baseline: Week 6, Week 30
Clinical: Remission in Disease Symptoms | Week 6, Week 30
  PCDAI ≤ 10: Week 6, Week 30
Clinical: Improvement in Serum Inflammatory Markers | Baseline, Week 6, Week 30
  Decrease C-reactive protein from baseline: Week 6, Week 30
Clinical: Improvement in Mucosal Inflammatory Markers | Baseline, Week 6, Week 30
  Decrease fecal calprotectin from baseline: Week 6, Week 30
Clinical: Change in Urine Metabolomics | Baseline, Week 6, Week 30
  Change in urine metabolite profile from baseline: Week 6, Week 30
Clinical: Change in Fecal Microbiome | Baseline, Week 6, Week 30
  Change in fecal 16s rRNA + metagenomics profile baseline: Week 6, Week 30

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Pai, BSc, CNSC, MD, FRCPC, Principal Investigator — McMaster Children's Hospital, Division of Pediatric Gastroenterology & Nutrition
Locations (2):
- Canada (2):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, University of Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Haberman Y, Tickle TL, Dexheimer PJ, Kim MO, Tang D, Karns R, Baldassano RN, Noe JD, Rosh J, Markowitz J, Heyman MB, Griffiths AM, Crandall WV, Mack DR, Baker SS, Huttenhower C, Keljo DJ, Hyams JS, Kugathasan S, Walters TD, Aronow B, Xavier RJ, Gevers D, Denson LA. Pediatric Crohn disease patients exhibit specific ileal transcriptome and microbiome signature. J Clin Invest. 2014 Aug;124(8):3617-33. doi: 10.1172/JCI75436. Epub 2014 Jul 8. PMID 25003194
- [Background] Gevers D, Kugathasan S, Denson LA, Vazquez-Baeza Y, Van Treuren W, Ren B, Schwager E, Knights D, Song SJ, Yassour M, Morgan XC, Kostic AD, Luo C, Gonzalez A, McDonald D, Haberman Y, Walters T, Baker S, Rosh J, Stephens M, Heyman M, Markowitz J, Baldassano R, Griffiths A, Sylvester F, Mack D, Kim S, Crandall W, Hyams J, Huttenhower C, Knight R, Xavier RJ. The treatment-naive microbiome in new-onset Crohn's disease. Cell Host Microbe. 2014 Mar 12;15(3):382-392. doi: 10.1016/j.chom.2014.02.005. PMID 24629344
- [Background] Maslowski KM, Vieira AT, Ng A, Kranich J, Sierro F, Yu D, Schilter HC, Rolph MS, Mackay F, Artis D, Xavier RJ, Teixeira MM, Mackay CR. Regulation of inflammatory responses by gut microbiota and chemoattractant receptor GPR43. Nature. 2009 Oct 29;461(7268):1282-6. doi: 10.1038/nature08530. PMID 19865172
- [Background] Conte MP, Schippa S, Zamboni I, Penta M, Chiarini F, Seganti L, Osborn J, Falconieri P, Borrelli O, Cucchiara S. Gut-associated bacterial microbiota in paediatric patients with inflammatory bowel disease. Gut. 2006 Dec;55(12):1760-7. doi: 10.1136/gut.2005.078824. Epub 2006 Apr 28. PMID 16648155
- [Background] Tedelind S, Westberg F, Kjerrulf M, Vidal A. Anti-inflammatory properties of the short-chain fatty acids acetate and propionate: a study with relevance to inflammatory bowel disease. World J Gastroenterol. 2007 May 28;13(20):2826-32. doi: 10.3748/wjg.v13.i20.2826. PMID 17569118
- [Background] Machiels K, Joossens M, Sabino J, De Preter V, Arijs I, Eeckhaut V, Ballet V, Claes K, Van Immerseel F, Verbeke K, Ferrante M, Verhaegen J, Rutgeerts P, Vermeire S. A decrease of the butyrate-producing species Roseburia hominis and Faecalibacterium prausnitzii defines dysbiosis in patients with ulcerative colitis. Gut. 2014 Aug;63(8):1275-83. doi: 10.1136/gutjnl-2013-304833. Epub 2013 Sep 10. PMID 24021287
- [Background] Sekirov I, Russell SL, Antunes LC, Finlay BB. Gut microbiota in health and disease. Physiol Rev. 2010 Jul;90(3):859-904. doi: 10.1152/physrev.00045.2009. PMID 20664075
- [Background] Putignani L, Del Chierico F, Petrucca A, Vernocchi P, Dallapiccola B. The human gut microbiota: a dynamic interplay with the host from birth to senescence settled during childhood. Pediatr Res. 2014 Jul;76(1):2-10. doi: 10.1038/pr.2014.49. Epub 2014 Apr 14. PMID 24732106
- [Background] Kunde S, Pham A, Bonczyk S, Crumb T, Duba M, Conrad H Jr, Cloney D, Kugathasan S. Safety, tolerability, and clinical response after fecal transplantation in children and young adults with ulcerative colitis. J Pediatr Gastroenterol Nutr. 2013 Jun;56(6):597-601. doi: 10.1097/MPG.0b013e318292fa0d. PMID 23542823
- [Background] Kellermayer R, Nagy-Szakal D, Harris RA, Luna RA, Pitashny M, Schady D, Mir SA, Lopez ME, Gilger MA, Belmont J, Hollister EB, Versalovic J. Serial fecal microbiota transplantation alters mucosal gene expression in pediatric ulcerative colitis. Am J Gastroenterol. 2015 Apr;110(4):604-6. doi: 10.1038/ajg.2015.19. No abstract available. PMID 25853207
- [Background] Suskind DL, Brittnacher MJ, Wahbeh G, Shaffer ML, Hayden HS, Qin X, Singh N, Damman CJ, Hager KR, Nielson H, Miller SI. Fecal microbial transplant effect on clinical outcomes and fecal microbiome in active Crohn's disease. Inflamm Bowel Dis. 2015 Mar;21(3):556-63. doi: 10.1097/MIB.0000000000000307. PMID 25647155
- [Background] Vandenplas Y, Veereman G, van der Werff Ten Bosch J, Goossens A, Pierard D, Samsom JN, Escher JC. Fecal Microbial Transplantation in Early-Onset Colitis: Caution Advised. J Pediatr Gastroenterol Nutr. 2015 Sep;61(3):e12-4. doi: 10.1097/MPG.0000000000000281. No abstract available. PMID 24399213
- [Background] Suskind DL, Singh N, Nielson H, Wahbeh G. Fecal microbial transplant via nasogastric tube for active pediatric ulcerative colitis. J Pediatr Gastroenterol Nutr. 2015 Jan;60(1):27-9. doi: 10.1097/MPG.0000000000000544. PMID 25162366
- [Background] Shimizu H, Arai K, Abe J, Nakabayashi K, Yoshioka T, Hosoi K, Kuroda M. Repeated fecal microbiota transplantation in a child with ulcerative colitis. Pediatr Int. 2016 Aug;58(8):781-5. doi: 10.1111/ped.12967. Epub 2016 Jun 21. PMID 27324973
- [Background] Turner D, Otley AR, Mack D, Hyams J, de Bruijne J, Uusoue K, Walters TD, Zachos M, Mamula P, Beaton DE, Steinhart AH, Griffiths AM. Development, validation, and evaluation of a pediatric ulcerative colitis activity index: a prospective multicenter study. Gastroenterology. 2007 Aug;133(2):423-32. doi: 10.1053/j.gastro.2007.05.029. Epub 2007 May 21. PMID 17681163
- [Background] Hyams JS, Ferry GD, Mandel FS, Gryboski JD, Kibort PM, Kirschner BS, Griffiths AM, Katz AJ, Grand RJ, Boyle JT, et al. Development and validation of a pediatric Crohn's disease activity index. J Pediatr Gastroenterol Nutr. 1991 May;12(4):439-47. PMID 1678008
- [Background] Pai N, Popov J. Protocol for a randomised, placebo-controlled pilot study for assessing feasibility and efficacy of faecal microbiota transplantation in a paediatric ulcerative colitis population: PediFETCh trial. BMJ Open. 2017 Aug 21;7(8):e016698. doi: 10.1136/bmjopen-2017-016698. PMID 28827258
- [Background] Orenstein R, Dubberke E, Hardi R, Ray A, Mullane K, Pardi DS, Ramesh MS; PUNCH CD Investigators. Safety and Durability of RBX2660 (Microbiota Suspension) for Recurrent Clostridium difficile Infection: Results of the PUNCH CD Study. Clin Infect Dis. 2016 Mar 1;62(5):596-602. doi: 10.1093/cid/civ938. Epub 2015 Nov 12. PMID 26565008
- [Background] Kelly CR, Ihunnah C, Fischer M, Khoruts A, Surawicz C, Afzali A, Aroniadis O, Barto A, Borody T, Giovanelli A, Gordon S, Gluck M, Hohmann EL, Kao D, Kao JY, McQuillen DP, Mellow M, Rank KM, Rao K, Ray A, Schwartz MA, Singh N, Stollman N, Suskind DL, Vindigni SM, Youngster I, Brandt L. Fecal microbiota transplant for treatment of Clostridium difficile infection in immunocompromised patients. Am J Gastroenterol. 2014 Jul;109(7):1065-71. doi: 10.1038/ajg.2014.133. Epub 2014 Jun 3. PMID 24890442
- [Background] Lobaton T, Bessissow T, De Hertogh G, Lemmens B, Maedler C, Van Assche G, Vermeire S, Bisschops R, Rutgeerts P, Bitton A, Afif W, Marcus V, Ferrante M. The Modified Mayo Endoscopic Score (MMES): A New Index for the Assessment of Extension and Severity of Endoscopic Activity in Ulcerative Colitis Patients. J Crohns Colitis. 2015 Oct;9(10):846-52. doi: 10.1093/ecco-jcc/jjv111. Epub 2015 Jun 26. PMID 26116558
- [Background] Cammarota G, Ianiro G, Tilg H, Rajilic-Stojanovic M, Kump P, Satokari R, Sokol H, Arkkila P, Pintus C, Hart A, Segal J, Aloi M, Masucci L, Molinaro A, Scaldaferri F, Gasbarrini G, Lopez-Sanroman A, Link A, de Groot P, de Vos WM, Hogenauer C, Malfertheiner P, Mattila E, Milosavljevic T, Nieuwdorp M, Sanguinetti M, Simren M, Gasbarrini A; European FMT Working Group. European consensus conference on faecal microbiota transplantation in clinical practice. Gut. 2017 Apr;66(4):569-580. doi: 10.1136/gutjnl-2016-313017. Epub 2017 Jan 13. PMID 28087657
- [Background] Agrawal M, Aroniadis OC, Brandt LJ, Kelly C, Freeman S, Surawicz C, Broussard E, Stollman N, Giovanelli A, Smith B, Yen E, Trivedi A, Hubble L, Kao D, Borody T, Finlayson S, Ray A, Smith R. The Long-term Efficacy and Safety of Fecal Microbiota Transplant for Recurrent, Severe, and Complicated Clostridium difficile Infection in 146 Elderly Individuals. J Clin Gastroenterol. 2016 May-Jun;50(5):403-7. doi: 10.1097/MCG.0000000000000410. PMID 26352106
- [Background] General Assembly of the World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. J Am Coll Dent. 2014 Summer;81(3):14-8. PMID 25951678
- [Derived] Pai N, Popov J, Hill L, Hartung E. Protocol for a double-blind, randomised, placebo-controlled pilot study for assessing the feasibility and efficacy of faecal microbiota transplant in a paediatric Crohn's disease population: PediCRaFT Trial. BMJ Open. 2019 Nov 28;9(11):e030120. doi: 10.1136/bmjopen-2019-030120. PMID 31784432